CLINICAL TRIAL: NCT05222789
Title: Postoperative Pain Assessment in Patients Undergoing Scheduled Laparoscopic Intestinal Resection Surgery
Brief Title: Postoperative Pain in Patients Undergoing Scheduled Laparoscopic Intestinal Resection Surgery
Acronym: TAP
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: ARP-ANA-2015-01
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain, Acute; Postoperative Pain, Chronic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TAP block: Patients receiving TAP block preoperatively, following routine clinical practice
  Interventions: Procedure: TAP
- Non-TAP: Patients not receiving TAP block preoperatively, following routine clinical practice

INTERVENTIONS:
Procedure: TAP — The transverse abdominal plane (TAP) block is a regional anesthesia technique performed using ultrasound that blocks the afferent nerves of the anterolateral abdominal wall, injecting local anesthetic in the fascial plane between the deep oblique and the transversus abdominis muscles.
  Groups: TAP block

SUMMARY:
This observational prospective study aims to evaluate the postoperative analgesic effect of a regional anesthesia thechnique (TAP block) in patients undergoing scheduled laparoscopic intestinal resection for intestinal cancer. ASA I-III patients operated between May 1 and September 30, 2019 under general anesthesia according to usual clinical practice, will be included. Patients who meet any of the following criteria will be excluded from this study: under 18 years old, language barrier, cognitive impairment or inability to assist in clinical assessment, drug or alcohol abuse, intake of opioids, consumption of analgesics 24 hours before surgery, BMI <18 or >35 kg/m2. Subsequently, an analysis will be made evaluating the quality of analgesia and the appearance of postoperative chronic pain and comparing the patients who underwent TAP block with those who did not.

DETAILED DESCRIPTION:
The transverse abdominal plane (TAP) block is a regional anesthesia technique that blocks the afferent nerves of the anterolateral abdominal wall. This observational prospective study aims to evaluate the postoperative analgesic effect in patients undergoing laparoscopic intestinal resection. ASA I-III patients operated on a scheduled basis, between May 1 and September 30, 2019, by laparoscopy for intestinal cancer resection under general anesthesia according to usual clinical practice, will be included. Patients who meet any of the following criteria will be excluded from this study: under 18 years old, language barrier, cognitive impairment or inability to assist in clinical assessment, drug or alcohol abuse, intake of opioids, consumption of analgesics 24 hours before surgery, BMI <18 or >35 kg/m2. Subsequently, an analysis will be made evaluating the quality of analgesia and the appearance of postoperative chronic pain and comparing the patients who underwent TAP block with those who did not.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Operated on a scheduled basis for laparoscopic intestinal cancer resection

Exclusion Criteria:

* Under 18 years old
* Language barrier
* Cognitive impairment or inability to collaborate in clinical assessment during the study
* Drug or alcohol abuse
* Habitual intake of opioids
* Consumption of analgesics 24 hours before surgery
* BMI <18 or >35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational prospective study comparing routine practice of analgesic management in consecutive surgical patients scheduled to undergo elective intestinal laparoscopic resection for suffering from intestinal cancer. 60 patients are expected to be included in this study and perioperative analgesic management prewarming will be performed following routine clinical practice. TAP block will be performed peroperatively under ultrasound control according to the anesthesiologist's decision. The patients will be followed up during the hospital stay (approximately one week) to evaluate the perioperative analgesic evolution and the appearance of secondary effects. A control will be carried out two years after surgery to evaluate the appearance of postoperative chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Postoperative acute pain assessed using Visual Analogue Scale, from 0 to 10 | from the arrival to the postanesthesia care unit to the 4 postoperative hours
  assessed using visual analogue scale
Intraoperative analgesic consumption | from the anesthesia induction to the end of the surgery
  assessed measuring the perioperative analgesics provided during the intraoperative period following routine clinical practice

SECONDARY OUTCOMES:
Postoperative chronic pain assessed using Visual Analogue Scale, from 0 to 10 | 2 years postoperatively
  assessed using visual analogue scale
Side effects | from the arrival to the postanesthesia care unit to the hospital discharge (7 days postoperatively)
  to record the perioperative side effects secondary to the analgesia administered perioperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Becerra, Principal Investigator — Hospital Universitario de Gran Canaria Doctor Negrín
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided